CLINICAL TRIAL: NCT02054923
Title: The Effect of Routine Video-recording on Colonoscopy Quality Indicators: a Cluster Randomized Trial.
Brief Title: The Effect of Routine Video-recording on Colonoscopy Quality Indicators.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other); Foundation for Polish Science (Unknown); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-QUALY
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer
Keywords: colonoscopy; videorecording; quality indicators; screening; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine video recording group (Experimental): Intervention: Procedure: Implementation of routine videorecording of colonoscopy withdrawal
  Interventions: Procedure: Implementation of routine videorecording
- Control group (Active Comparator): Intervention: Behavioral: No routine videorecording (on demand videorecording possible)
  Interventions: Behavioral: No routine videorecording

INTERVENTIONS:
Procedure: Implementation of routine videorecording — All screening centres (clusters) assigned to the routine video recording group will receive an appropriate number of video recorders and DVDs for each colonoscopy room. Screening centre coordinators will be responsible for the implementation of routine video recording of all screening colonoscopies (only withdrawal) in the centres. Every three months screening centre coordinators will be asked to send back all recorded DVDs. All the recorded DVDs will be reviewed to verify ceacal intubation and withdrawal time by the PCSP team and then stored.
  Arms: Routine video recording group
Behavioral: No routine videorecording — Screening centres (clusters) assigned to the control group will not receive video recorders and DVDs but will be allowed to record colonoscopies on demand.
  Arms: Control group

SUMMARY:
Routine video recording of the colonoscopy examination has been proposed as a simple and easy to implement method that could improve the quality of colonoscopy. The purpose of this study is to investigate whether implementation of routine video recording of screening colonoscopy withdrawal is effective as a means of supporting quality performance of colonoscopy. The study will be performed in 8 screening centers within the framework of a national colonoscopy screening program in Poland (the Polish Colonoscopy Screening Platform; PCSP). Individuals aged 55-64 years are eligible to participate in the PCSP. In the run-in period colonoscopy quality measures will be monitored through a dedicated joint database. Then eligible screening centres will be randomly assigned in a 1:1 ratio to the video recording group or the control group. Screening centres assigned to the video recording group will receive videorecorders and DVDs and will be asked to video record all screening colonoscopies (only withdrawal). Control group will be allowed to record colonoscopies on demand only. Then , the colonoscopy quality measures will again be monitored through a dedicated joint database. All the recorded DVDs will be reviewed to verify ceacal intubation and withdrawal time by the PCSP team.

ELIGIBILITY:
Inclusion Criteria:

* Screening centres participating in the Polish Colonoscopy Screening Platform (PCSP) between 2012 and 2013, in which no routine video recording of screening colonoscopies is performed
* Screening centres which will sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5200 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in screening centre adenoma detection rate before and after intervention | From the time of randomization up to 10 months (the end of screening program annual edition)
  Proportion of patients with at least one adenoma identified (measured in screening program database).

SECONDARY OUTCOMES:
Reported and audited ceacal intubation rates | From the time of randomization up to 10 months (the end of screening program annual edition)
  Proportion of complete colonoscopies (measured in screening program database; audited ceacal intubation rates will be assessed through videorecording review)
Rates of painful colonoscopy | From the time of randomization up to 10 months (the end of screening program annual edition)
  Severe or moderate pain on a four point verbal rating scale (measured in screening program database)
Rates of proximal (to the splenic flexure) serrated polyps ≥10mm in size | From the time of randomization up to 10 months (the end of screening program annual edition)
  Measured in screening program database.

CONTACTS AND LOCATIONS:
Overall Officials: Michal F. Kaminski, MD, PhD, Principal Investigator — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology; Jaroslaw Regula, MD, PhD, Study Chair — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland; Maria Rupińska, Study Director — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology, Warsaw, Poland